CLINICAL TRIAL: NCT03798600
Title: Pharmacokinetics/Pharmacodynamics (PK/PD) of Caspofungin in Intensive Care Unit (ICU) Patients. An Open Observational Study for Antifungal Treatment's Optimization
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, Principal investigator, Careggi Hospital
Other Study IDs: CEAVC, 32366/2015; OSS.15.114
Record Dates: First submitted 2019-01-04; First posted 2019-01-10 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Critical Illness; Infection
Keywords: Caspofungin; pharmacokinetic; pharmacodynamic
MeSH Terms: conditions — Critical Illness; Infections | interventions — Caspofungin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine samples. To perform the PK study, blood samples (of approximately 2 ml each) will be obtained at different time points following the first administration. These samples will occur at the same time of routine blood gas analysis (hourly obtained in the ICU) and no further extra-routine blood samples will be required for this study. In particular, the blood that normally remains in the syringe of blood gas analysis, and usually thrown as waste fluid, will be saved and used for PK analysis. Thus, no increase in blood sampling from the patient will be obtained, both in terms of frequency of sampling or volume of blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically ill patients: 20 patients consecutively admitted in the ICU with severe sepsis or septic shock requiring caspofungin therapy will be considered for this observational study.
  Inclusion Criteria:
  Adult ICU patients (>18 yrs) with severe sepsis or septic shock undergoing caspofungin therapy based on clinical judgement (empiric therapy) or microbiological result (targeted therapy).
  Exclusion criteria:
  Concomitant ciclosporin or rifampicin therapy. Pregnancy Continuous renal replacement therapy Severe Liver failure (Child Pugh score > 6)
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — In accordance with routine clinical practice, Caspofungin will be given at the loading dose of 70 mg followed by 50 mg daily (for people < 80 kg body weight). No dose reduction will be performed in Child-Pugh score A or B. Duration of therapy will be performed in accordance with ESCMID guidelines and clinical conditions.

SUMMARY:
PK of Caspofungin in ICU septic patients might be changed as compared to healthy volunteers due to sepsis-related pathophysiology.

Sub-optimal plasma and tissue concentrations might be achieved in these patients when drugs are administered at the same dosage/regimen suggested for healthy volunteers.

DETAILED DESCRIPTION:
Open non randomized, non controlled single center study on the pharmacokinetics of caspofungin in 20 consecutive ICU patients with severe sepsis or septic shock, requiring caspofungin therapy and PK-PD evaluation for the optimization of caspofungin therapy. The aim of this study is to describe the Caspofungin PK-PD alterations in a cohort of critically ill septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients (>18 yrs)
* Severe sepsis or septic shock
* Caspofungin therapy based on clinical judgement (empiric therapy) or microbiological result (targeted therapy).

Exclusion Criteria:

* Concomitant ciclosporin or rifampicin therapy.
* Pregnancy
* Continuous renal replacement therapy
* Severe Liver failure (Child Pugh score > 6)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 20 patients consecutively admitted in the ICU with severe sepsis or septic shock requiring caspofungin therapy will be considered for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Alterations of Caspofungin Area Under the curve (AUC) in septic patients admitted to the Intensive Care Unit (ICU). | first 24 hours after loading dose
  The caspofungin AUC will be described and compared with that reported in the literature for healthy volunteers.

SECONDARY OUTCOMES:
Alterations of Cmax/MIC target - which guarantees the maximal exposure of Candida spp to caspofungin | first 24 hours after loading dose
  The Cmax/MIC ratio, will be calculated and compared with that reported in the literature to obtain the infection eradication.
Alterations of Cmax/MIC target - which guarantees the maximal exposure of Candida spp to caspofungin | at day 4 after loading dose
  The Cmax/MIC ratio, will be calculated and compared with that reported in the literature to obtain the infection eradication.
Alterations of AUC/MIC target - which guarantees the maximal exposure of Candida spp to caspofungin | first 24 hours after loading dose
  The AUC/MIC ratio, will be calculated and compared with that reported in the literature to obtain the infection eradication.
Alterations of AUC/MIC target - which guarantees the maximal exposure of Candida spp to caspofungin | at day 4 after loading dose
  The AUC/MIC ratio, will be calculated and compared with that reported in the literature to obtain the infection eradication.
Alterations of Caspofungin maximum serum concentrations in septic patients admitted to the Intensive Care Unit (ICU). | first 24 hours after loading dose
  The caspofungin maximum serum concentrations will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin maximum serum concentrations in septic patients admitted to the Intensive Care Unit (ICU). | at day 4 after loading dose
  The caspofungin maximum serum concentrations will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin minimum serum concentrations in septic patients admitted to the Intensive Care Unit (ICU). | first 24 hours after loading dose
  The caspofungin minimum serum concentrations will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin minimum serum concentrations in septic patients admitted to the Intensive Care Unit (ICU). | at day 4 after loading dose
  The caspofungin minimum serum concentrations will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin volume distribution in septic patients admitted to the Intensive Care Unit (ICU). | first 24 hours after loading dose
  The caspofungin volume distribution will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin volume distribution in septic patients admitted to the Intensive Care Unit (ICU). | at day 4 after loading dose
  The caspofungin volume distribution will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin elimination half life in septic patients admitted to the Intensive Care Unit (ICU). | first 24 hours after loading dose
  The caspofungin elimination half life will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin elimination half life in septic patients admitted to the Intensive Care Unit (ICU). | at day 4 after loading dose
  The caspofungin elimination half life will be described and compared with those reported in the literature for healthy volunteers.
Alterations of Caspofungin Area Under the curve (AUC) in septic patients admitted to the Intensive Care Unit (ICU). | at day 4 after loading dose
  The caspofungin AUC will be described and compared with that reported in the literature for healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Villa, MD, Principal Investigator — Azienda Careggi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adembri C, Villa G, Rosi E, Tofani L, Fallani S, De Gaudio AR, Novelli A. Caspofungin PK in critically ill patients after the first and fourth doses: suggestions for therapeutic drug monitoring? J Chemother. 2020 May;32(3):124-131. doi: 10.1080/1120009X.2020.1737783. Epub 2020 Mar 23. PMID 32202224